CLINICAL TRIAL: NCT02248987
Title: Study on Abnormal Dopamine Synthesis and Connectivity According to the Antipsychotic Treatment Response in Schizophrenia
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jun Soo Kwon, professor, Seoul National University Hospital
Other Study IDs: 3420130030
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Antipsychotic Agents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Clozapine: stable patients treated with clozapine
  Interventions: Other: patients treated with antipsychotics
- Other antipsychotics: stable patients treated with risperidone or paliperidone or olanzapine
  Interventions: Other: patients treated with antipsychotics
- Healthy volunteer: healthy controls
  Interventions: Other: patients treated with antipsychotics

INTERVENTIONS:
Other: patients treated with antipsychotics

SUMMARY:
The purpose of this study is to evaluate abnormal dopamine synthesis and connectivity according to the antipsychotic treatment response in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia
* clinically stable state

Exclusion Criteria:

* history of previous head injury, epileptic disorder, other medical comorbidity
* substance abuse/dependence

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Schizophrenia patients treated with clozapine
  2. Schizophrenia patients treated with risperidone or paliperidone or olanzapine
  3. Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Striatal [18F]-DOPA uptake measured using positron emission tomographic 18F-dopa imaging. | within 2 weeks from enrollment

SECONDARY OUTCOMES:
resting state functional magnetic resonance imaging | within 2 weeks from enrollment
diffusion tensor imaging | within 2 weeks from enrollment
clinical measure including Positive and Negative Syndrome Scale | within 2 weeks from enrollment
neurocognitive function test | within 2 weeks from enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea